CLINICAL TRIAL: NCT03572088
Title: Terlipressin Infusion During Whipple Procedure: Effect on Blood Loss and Transfusion Needs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magdy Mohammed Mahdy Sayed, Assiut-Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABC-223-DE
Record Dates: First submitted 2018-06-17; First posted 2018-06-28 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Terlipressin; Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Terlipressin; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Terlipresssin (Active Comparator): Terlipressin was started at the beginning of surgery, just after exposure of the portal vein and getting a basal portal pressure reading, as an initial bolus dose of 1 mg over 30 minutes (1 mg/50 ml normal saline at a rate of 100 ml/h) followed by a continuous infusion of 2 μg/kg/h(1 mg/50 ml at a rate equal to wt/10 ml per hour) and weaned in the postoperative period over 4 hours.
  Interventions: Drug: Terlipressin
- Control (Placebo Comparator): patients received the same volume of normal saline for the same duration (50 ml normal saline at a rate of 100 ml/h followed by a continuous infusion of 50 ml at a rate equal to wt/10 ml per hour and weaned in the postoperative period over 4 hours)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Terlipressin — Terlipressin is a synthetic vasopressin analogue with relative specificity for the splanchnic circulation(Terlipressin was started at the beginning of surgery as an initial bolus dose of 1 mg over 30 mints(1 mg/50 ml normal saline at a rate of 100 ml/h) followed by a continuous infusion of 2 μg/kg/h(1 mg/50 ml at a rate equal to wt/10 ml per hour) and weaned in the postoperative period over 4 hours.)
  Other Names: glypressin
  Arms: Terlipresssin
Drug: normal saline — Patients received 50 ml normal saline at a rate of 100 ml/h followed by a continuous infusion of 50 ml at a rate equal to wt/10 ml per hour and weaned in the postoperative period over 4 hours.
  Other Names: 0.9 Nacl
  Arms: Control

SUMMARY:
The present study aims to look at the effect of terlipressin infusion on blood loss and blood transfusion needs during Whipple procedure

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of age,
* ASA classification class I and II,
* Patients assigned for Whipple procedure.

Exclusion Criteria:

* Preoperative renal failure,
* Severe liver dysfunction (Child-Turcotte-Pugh grade C),
* Hyponatremia (Na+ <132mmol/l),
* Severe valvular heart disease,
* Heart failure,
* Symptomatic coronary heart disease,
* Bradycardic arrhythmia (heart rate < 60/min),
* Peripheral artery occlusive disease (clinical stadium II-IV),
* Uncontrolled arterial hypertension (Blood pressure >160/100mmHg despite intensive treatment),
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | intaoperative periods
  Amount of intraoperative blood loss in ml

SECONDARY OUTCOMES:
Patients needing blood transfusion | intaoperative periods
  Number of patients needing blood transfusion
Red blood cell units transfused | intaoperative periods
  The number of red blood cell units transfused
portal pressure changes | intaoperative periods
  portal pressure changes in mmHg
ICU stay | postoperative periods
  ICU stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Assiut University hospital Egypt, Egypt, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided